CLINICAL TRIAL: NCT02548169
Title: A Phase I, Safety Trial of Dendritic Cell Vaccine and Chemotherapy for Patients With Pancreatic Cancer
Brief Title: Dendritic Cell Vaccine and Chemotherapy for Patients With Pancreatic Cancer
Acronym: PancVax
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped because of loss of funding and no safety issues
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015-119
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
Keywords: Dendritic Cell Vaccine; FOLFIRINOX; nab-paclitaxel; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Group 1 will consist of patients with resectable, borderline resectable or locally advanced pancreatic cancer. Group 1 will receive DC Vaccine + Standard of Care Chemotherapy.
  Interventions: Biological: DC Vaccine + Standard of Care Chemotherapy
- Group 2 (Active Comparator): Group 2 will consist of patients with metastatic pancreatic cancer, newly diagnosed/untreated metastatic pancreatic cancer, or metastatic pancreatic cancer who have undergone prior neo-adjuvant therapy. Group 2 will receive DC Vaccine + Standard of Care Chemotherapy.
  Interventions: Biological: DC Vaccine + Standard of Care Chemotherapy

INTERVENTIONS:
Biological: DC Vaccine + Standard of Care Chemotherapy — 4 doses of DC vaccine at 2 weeks interval, combined with either:
  * Standard of care neoadjuvant folinic acid, oxaliplatin, irinotecan and 5- Fluorouracil (5FU) (FOLFIRINOX) regimen alone (6 cycles)
  * FOLRIRINOX regimen followed by 5-FU chemoradiation or Gemcitabine Chemoradiation
  * Gemcitabine + nab-paclitaxel
  The first vaccination will include one intradermal injection of 100 μL at 15 x106 cells/mL in the upper thigh and one subcutaneous injection of 1 mL (15 x 106 cells/mL) .
  The participants will receive 3 additional subcutaneous vaccinations, each injection of 1 mL at 15 x 106 cells/mL, at 2 weeks interval, on Day 2 of study weeks 3, 5 and 7.
  Participants will receive 2 booster DC vaccinations subcutaneously of 1 mL at 15x106 cells/mL.

SUMMARY:
The primary objective is to confirm clinical safety and feasibility of combining the antigen-loaded Dendritic Cell (DC) vaccine with chemotherapy including folinic acid, oxaliplatin, irinotecan and 5-Fluorouracil (5FU) (FOLFIRINOX) and nab-paclitaxel/gemcitabine in patients with pancreatic cancer.

The secondary objectives of this trial are to determine preliminary clinical efficacy based on response rates, overall survival and progression free survival compared with historic control, and surgical conversion rate as defined as percent of locally advanced (unresectable) patients achieving resectability within 6 months of treatment initiation. Also, to identify vaccine immunogenicity by measuring acquired, T cell-mediated immune activating events post-vaccination and to correlate clinical response with acquired immune responses.

DETAILED DESCRIPTION:
This is a single center, exploratory pilot safety, open label, phase I trial that will evaluate the combination of DC vaccination in 2 groups of patients when combined with chemotherapy including FOLFIRINOX and gemcitabine+nab-paclitaxel in patients with pancreatic cancer. The investigations will accrue 20 evaluable subjects over 20 months with 10 patients in each group. Subjects will be assigned to group 1 or group 2 according to the subject's disease stage.

The protocol will be conducted in two stages:

The 1st 3 patients will be enrolled to either group to receive DC vaccinations combined with standard chemotherapy. A safety analysis will be performed after the first 3 patients have completed 6 vaccines. If no vaccine dose-limiting toxicity occurs in any of the 3 patients then the study will proceed with stage 2. Stage 2 will include the enrollment of the remaining 17 patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected pancreatic ductal adenocarcinoma (PDAC) prior to diagnosis or histological diagnosis of adenocarcinoma of the pancreas confirmed by pathology.
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.
* Serum Albumin greater than or equal to 2.0 gm/dL
* Expected survival greater than or equal to 6 months.
* Adequate hematologic function as defined by
* Absolute Neutrophil Count (ANC) greater than 1500/mm^3
* Platelets greater than or equal to 70,000/mm^3
* Hemoglobin greater than 9 g/dL
* Adequate liver function, as defined by:
* Serum Total Bilirubin less than or equal to 2 x Upper limit of normal (ULN) mg/dL
* Alanine transaminase (ALT) and Aspartate transaminase (AST) less than or equal to 2.5x Upper limit of normal (ULN)
* Serum Creatinine less than or equal to 2 x Upper limit of normal (ULN) or creatinine clearance greater than or equal to 30 ml/min
* All females of child bearing potential must agree to use contraception to avoid pregnancy throughout the study and for 1 month after the last DC vaccination.
* Subjects must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate. Subjects may not be consented by a medical power of attorney.
* Subject must be accessible for treatment and follow up.

Exclusion Criteria:

* History of Organ transplant
* Other malignancy within 5 years, unless the probability of recurrence of the prior malignancy is <5% as determined by the principal investigator.
* Current, active immunosuppressive therapy such as cyclosporine, tacrolimus
* Subjects taking chronic systemic corticosteroid therapy for any reason are not eligible. Subjects may receive steroids as prophylactic anti-emetics, not toe exceed 10mg Decadron weekly. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require chronic systemic corticosteroids after beginning vaccination will be removed from the study.
* Significant or uncontrolled congestive heart failure, myocardial infarction or significant ventricular arrhythmias within the last 6 months
* Active infection or antibiotics within 48 hours prior to study enrollment, including unexplained fever
* Autoimmune disease ( e.g. systemic lupus erythematosis, rheumatoid arthritis). Subjects with remote history of asthma or mild active asthma are eligible.
* Other severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as:
* Severe impaired lung functions as defined by spirometry and diffusing capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
* Uncontrolled diabetes as defined by fasting serum glucose >250 mg/dL
* Live disease such as cirrhosis or severe hepatic impairment (child pugh class C)
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or quality of the data.
* Other investigational or anti-cancer treatments while participating in this study.
* Other active cancer
* Women who are pregnant or breastfeeding
* Known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of combining the DC vaccine with chemotherapy DC vaccine dose-limiting toxicities will be measured according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 | 3 Years
  Follow up for toxicity will be recorded for the first 30 days following the last DC vaccination and any long-term toxicity will be followed for 3 years after completing study therapy.

SECONDARY OUTCOMES:
Objective Response | 3 years
  Overall response rate will be assessed by using standard Response Evaluation Criteria in Solid Tumors (RECIST).
Overall Survival | 3 years
  Time from the start of therapy to death from any cause.
Progression Free Survival | 3 Years
  Time from enrollment until objective tumor progression or death
Average of all changes in Quality of Life (QoL) Score | 3 Years
  Quality of Life score will be assessed by using self-administered questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Becerra, MD, Principal Investigator — Charles A. Sammons Cancer Center/Texas Oncology
Locations (1):
- Charles A. Sammons Cancer Center, Dallas, Texas, United States